CLINICAL TRIAL: NCT06084390
Title: Interdisciplinary Rehabilitation for Patients With Chronic Pain in Primary Healthcare
Brief Title: Interdisciplinary Rehabilitation for Chronic Pain in Primary Healthcare
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Painteam
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain; Pain Management
Keywords: randomised controlled trial; primary care
MeSH Terms: conditions — Chronic Pain; Agnosia | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interdisciplinary rehabilitation + booster-session (intervention) (Experimental): Standard care by the interdisciplinary rehabilitation teams in primary healthcare + extended access to the team and a booster visit after 3 months.
  Interventions: Other: Interdisciplinary care + booster session (intervention)
- Interdisciplinary rehabilitation (control) (Active Comparator): Standard care by the interdisciplinary rehabilitation teams in primary healthcare.
  Interventions: Other: Interdisciplinary care (control)

INTERVENTIONS:
Other: Interdisciplinary care + booster session (intervention) — Standard care for interdisciplinary rehabilitation at any of the six interdisciplinary teams in primary health care in Region Västra Götaland, Sweden + one extra booster-session 3 months after the standard care rehabilitation. At the booster-session, the participant´s individual rehabilitation plan is followed-up and adjusted. This extra period also includes extended access to the team, meaning that the participants have the possibility to contact the team and, if needed, have digital or telephone contact.
  Arms: Interdisciplinary rehabilitation + booster-session (intervention)
Other: Interdisciplinary care (control) — Standard care for interdisciplinary rehabilitation at any of the six interdisciplinary teams in primary health care in Region Västra Götaland, Sweden.
  Arms: Interdisciplinary rehabilitation (control)

SUMMARY:
Purpose: The overall aim is to investigate the effect of interdisciplinary rehabilitation in primary health care (PHC) for patients with chronic pain. Specific questions: What is the effect of extended access to the interdisciplinary PHC pain team + a booster session after finishing the rehabilitation program? Does participation in PHC interdisciplinary rehabilitation contribute to health improvements and are there predictors of this? Method: A randomized controlled trial (RCT). 200 patients with chronic pain that participate in interdisciplinary rehabilitation in primary healthcare in Region Västra Götaland (VGR) in Sweden will be included in the RCT and randomized to Intervention; standard care by the interdisciplinary teams in PHC + extended access to the team and a booster session 3 months after the end of the rehabilitation, or Control; only standard care by the interdisciplinary teams. Outcomes are health related quality of life, pain intensity and other health aspects.

DETAILED DESCRIPTION:
The participants will be randomly allocated to intervention or active control. All participants in both arms receive the standard care for interdisciplinary rehabilitation at any of the six PHC pain teams in VGR. The teams consist of a physician, physiotherapist, occupational therapist and psychologist. All teams provide person-centred rehabilitation, aiming to increase physical activity and support behavioural changes, and to decrease symptoms and the impact of pain on the patients´ daily lives. The standard care interdisciplinary rehabilitation period contains both theoretical and practical components such as patient education, physical exercise and behavioural interventions. The sessions are mainly group-based. The duration of the rehabilitation period varies between 5 to 7 weeks + a follow-up visit after 3 months.

The participants in the intervention arm also receive an extra booster-session 3 months after the standard follow-up. At the booster-session, the participant´s individual rehabilitation plan is followed-up and adjusted. This extra period also includes extended access to the team, meaning that the participants have the possibility to contact the team and, if needed, have digital or telephone contact.

The participants complete a battery of questionaires included in the Swedish Quality Registry for Pain Rehabilitation an also extra questionnaires provided to the participants through an electronic research form.

Data collection is made at baseline before starting the rehabilitation, directly after the 5 to 7 weeks rehabilitation period and 6, 12 and 24 months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Persons participating in interdisciplinary team rehabilitation in primary healthcare in Region Västra Götaland, Sweden.

Exclusion Criteria:

* Severe psychiatric disease, language difficulties that makes it impossible to complete the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline, directly after the rehabilitation period and 6, 12 and 24 months from the end of the rehabilitation period.
  Assessed with visual analog scale and numeric rating scale (0-100 mm, higher is more severe pain)
Health related quality of life | Baseline, directly after the rehabilitation period and 6, 12 and 24 months from the end of the rehabilitation period.
  Rand-36 (0-100, a higher score indicates better health-related quality of life)
Health related quality of life 2 | Baseline, directly after the rehabilitation period and 6, 12 and 24 months from the end of the rehabilitation period.
  EuroQol 5D-3L (0-100, a higher score indicates better health-related quality of life)
Health related quality of life 3 | Baseline, directly after the rehabilitation period and 6, 12 and 24 months from the end of the rehabilitation period.
  EuroQol-Visual analogue scale (0-100, a higher score indicates better health-related quality of life)

SECONDARY OUTCOMES:
Pain spread | Baseline, directly after the rehabilitation period and 6, 12 and 24 months from the end of the rehabilitation period.
  The participants mark in boxes painful areas
Pain acceptance | Baseline, directly after the rehabilitation period and 6, 12 and 24 months from the end of the rehabilitation period.
  The Chronic pain acceptance questionnaire (CPAQ-8) (Total score 0-48, 2 subscales 0-24 p. Higher score means better pain acceptance)
Self-efficacy | Baseline, directly after the rehabilitation period and 6, 12 and 24 months from from the end of the rehabilitation period.
  The Pain self-efficacy questionnaire short-form (PSEQ_2) (0-12, a higher score means better self-efficacy)
Symptoms of stress | Baseline, directly after the rehabilitation period and 6, 12 and 24 months from the end of the rehabilitation period.
  The stress and crisis inventory (SCI-93) (0-140, a higher score means more stress) symptoms)
Physical activity | Baseline, directly after the rehabilitation period and 6, 12 and 24 months from the end of the rehabilitation period.
  The Godin questionnaire (hours of physical activity per week)
Anxiety and depression | Baseline, directly after the rehabilitation period and 6, 12 and 24 months from the end of the rehabilitation period.
  The hospital anxiety and depression scale (2 subscales for symptoms of anxiety and depression ranging from 0 to 21, a higher value means a higher degree of anxiety or depression)
Self-rated function | Baseline, directly after the rehabilitation period and 6, 12 and 24 months from the end of the rehabilitation period.
  The Functional rating index (0-100 %, higher percent is worse)
Work ability | Baseline, directly after the rehabilitation period and 6, 12 and 24 months from the end of the rehabilitation period.
  One question (number 7) from the Work ability index (0-10, higher score is better)
Life satisfaction | Baseline, directly after the rehabilitation period and 6, 12 and 24 months from the end of the rehabilitation period.
  The LiSat questionnaire (2 questions ranging 1-6, higher score is better life satisfaction)
Fatigue | Baseline, directly after the rehabilitation period and 6, 12 and 24 months from the end of the rehabilitation period.
  The multidimensional fatigue inventory (5 subscales ranging from 4 -20, higher score means more fatigue)
Pain catastrophizing | Baseline, directly after the rehabilitation period and 6, 12 and 24 months from the end of the rehabilitation period.
  The pain catastrophizing scale (Total score 0-52, higher score is worse)
Patients´ own impression of change | Directly after the rehabilitation period and 6, 12 and 24 months from the end of the rehabilitation period.
  Patient global impression of change (1-7, lower score means more improvement)
Health care use | From 12 months before to 24 months after the rehabilitation period.
  Health care visit statistics
Sickness abscence | From 12 months before to 24 months after the rehabilitation period.
  Sickness absence data

CONTACTS AND LOCATIONS:
Overall Officials: Anna Bergenheim, Dr, Principal Investigator — Research and development primary healthcare Fyrbodal, region Västra Götaland, Sweden
Locations (1):
- Research and development primary health care Fyrbodal, Vänersborg, Region Västra Götaland, Sweden

IPD SHARING:
Plan to Share IPD: No